CLINICAL TRIAL: NCT02392897
Title: Eating Frequency and Its Influence on Satiety and Biomarkers of Health & Disease
Brief Title: theFRESHstudy: FRequency of Eating and Its Influence on Satiety and Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 8292; 1R01DK103674-01 (NIH)
Record Dates: First submitted 2015-03-04; First posted 2015-03-19 (Estimated); Last update posted 2019-07-25 (Actual); Status verified 2019-07

CONDITIONS: Healthy
Keywords: meal frequency; eating frequency; ingestive frequency; Positive energy balance; Satiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- High Eating Frequency (Experimental): 6 Eating Occasions
  Interventions: Behavioral: High Eating Frequency
- Low Eating Frequency (Experimental): 3 Eating Occasions
  Interventions: Behavioral: Low Eating Frequency

INTERVENTIONS:
Behavioral: High Eating Frequency — Free-living participants will complete a 21-day high eating frequency (high EF) Phase in which consume all daily energy at 6 eating occasions.
  Arms: High Eating Frequency
Behavioral: Low Eating Frequency — Free-living participants will complete a 21-day low eating frequency (low EF) Phase
  Arms: Low Eating Frequency

SUMMARY:
Eating frequency may play an independent role in appetite regulation, overall caloric consumption and measures of long-term health or disease risk. Some literature recommends frequent eating, but pilot data suggest that this type of eating pattern may be harmful to health since it leaves the body in a perpetual fed state and increases systemic inflammation. Therefore, the investigators will conduct a clinical trial in 50 healthy adults to compare a low frequency eating pattern to a high frequency eating pattern in relation to blood-based markers of inflammation, metabolic health and appetite. Study results will be applied to recommendations for eating frequency in the context of an overall healthy diet.

DETAILED DESCRIPTION:
This proposal will investigate whether eating frequency influences health. Evidence-based recommendations are lacking for the optimal number of daily eating occasions. This is an important area of research because over the past 40 years Americans' eating habits have changed from three meals a day to a pattern whereby most people now have 6-8 daily eating occasions. Apart from potential increases in total energy intake, frequent eating leaves people in a constant postprandial state. This constant, modestly elevated glycemia disturbs the normal glucose-insulin and counter-regulatory hormone network balance and also disturbs downstream cell signaling pathways. A constant postprandial state may increase systemic inflammation and cause numerous other metabolic disturbances. As a result, eating frequency (EF) may be associated with risk of diet-related chronic diseases such as cardiovascular disease, cancer and diabetes, which are the major causes of morbidity, mortality and health care costs in the U.S. To better understand this phenomena the investigators propose a randomized, cross-over clinical trial to test a low-EF eating pattern (three eating occasions/day) vs. a high-EF eating pattern (six eating occasions/day) in relation to inflammation, an adipokine and appetite. The investigators hypothesize that compared to eating three times/day, eating six times/day will increase biomarkers of systemic inflammation, will decrease a beneficial adipokine and will increase both biomarkers and self-reported measures of appetite. The investigators will test their hypothesis with these specific aims: 1) To test the effects of low vs. high eating frequency on inflammatory biomarkers (fasting high-sensitivity C-reactive protein, Interleukin-6 and tumor necrosis factor-α,) and a beneficial adipokine (adiponectin); 2) To test the effects of low vs. high eating frequency on appetite [daily ratings of perceived appetite and serial ratings during a six-hour appetite testing session] and biomarkers involved in appetite regulation and food intake (leptin, ghrelin, peptide YY, and cholecystokinin). The investigators will enroll n=50 males and females who are normal weight, overweight or obese. Participants will complete two 3-week long isocaloric intervention periods in random order [low EF (three eating occasions/day) and high EF (six eating occasions/day)]. Participants will be free-living and eating their own food using study-provided structured meals plans. Study staff will provide on-going support and instruction to maximize adherence to the protocol. Fasting blood samples will be collected at the beginning and end of each study phase. The investigators will test for the intervention effect by using the GEE modification of linear regression to compare mean biomarker response (intervention effect) for each study phase. On the last day of each intervention period, participants will complete 6-hour appetite testing sessions where two test meals will be provided in the low-EF phase and four test meals will be provided in the high-EF phase. Serial appetite ratings and bloods will be collected to assess perceived appetite and hormones of appetite and satiety. Results from this investigation will be used to form guidelines for eating frequency in the context of an overall healthy diet.

ELIGIBILITY:
Inclusion Criteria:

* Normal, overweight and obese males and females
* BMI = 18.5-24.9 and 28.0-40.0 kg/m²
* Ages 18-50 years
* Live in Seattle, WA

Exclusion Criteria:

* Pregnant women
* Presence of diseases requiring dietary modification, including physician diagnosed cardiovascular disease or diabetes mellitus, use of medications that may impact study results including non-steroidal anti-inflammatory drugs (NSAIDS)
* Abnormal fasting glucose (>100 mg/dL)
* History of disordered or restrained eating and severe food restrictions
* Individuals with BMI ≥ 40 kg/m2

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2015-04; Primary Completion 2018-12-19 (Actual); Study Completion 2018-12-19 (Actual)

PRIMARY OUTCOMES:
Test the effects of low vs. high eating frequency on inflammatory biomarkers | 3 weeks
  To test the effects of low vs. high eating frequency on inflammatory biomarkers.

SECONDARY OUTCOMES:
Test the effects of low vs. high eating frequency on appetite | 3 weeks
  To test the effects of low vs. high eating frequency on subjective appetite as measured by visual analog scale
Test the effects of low vs. high eating frequency on appetite | 6 hours
  To test the effects of low vs. high eating frequency as measured by serial measures of appetite-related biomarkers

CONTACTS AND LOCATIONS:
Overall Officials: Marian Neuhouser, PhD, Principal Investigator — Fred Hutchinson Cancer Center
Locations (1):
- Fred Hutchinson Cancer Research Center, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhang X, Schenk JM, Perrigue M, Drewnowski A, Wang CY, Beatty SJ, Neuhouser ML. No Effect of High Eating Frequency Compared with Low Eating Frequency on Appetite and Inflammation Biomarkers: Results from a Randomized Crossover Clinical Trial. J Nutr. 2024 Aug;154(8):2422-2430. doi: 10.1016/j.tjnut.2024.04.029. Epub 2024 May 3. PMID 38703890